CLINICAL TRIAL: NCT00810589
Title: A Randomised, Single Centre, Double-Blind, Two-Period Crossover, Glucose Clamp Trial to Compare the Pharmacodynamic Effects of Single Doses of Insulin Detemir and Neutral Protamin Lispro (NPL) Insulin in Subjects With Type 1 Diabetes
Brief Title: A Randomised, Single Centre, Double-Blind, Two-Period Crossover, Glucose Clamp Trial
Acronym: ENM-HS-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Univ. Prof. Dr. Thomas Pieber, Medical University Graz, Internal Medicine, Endocrinology and Nuclear Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ENM-HS-001
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes, Type I
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Levemir
- 2 (Active Comparator)
  Interventions: Drug: Humalog NPL Insulin

INTERVENTIONS:
Drug: Levemir — 0,4 IE per kg bodyweight
  Other Names: Insulin Detemir
  Arms: 1
Drug: Humalog NPL Insulin — 0,4 IE per kg bodyweight
  Other Names: Humalog NPL
  Arms: 2

SUMMARY:
Clinical pharmacology trials investigating insulin detemir in subjects with type 1 diabetes have shown a prolonged and reproducible action profile of insulin detemir compared with NPH insulin and insulin glargine. Duration of action of insulin detemir has been reported to be up to 24 hours.9,10,11 It has, however, been proposed that the mean duration of action is underestimated in glucose clamps lasting only 24 hours. This is so because a duration of action longer than 24 hours in individual clamps will be set to 24 hours in the mean calculation, whereas a shorter duration of action in individual clamps will be set to the true value.

It has been shown in clinical pharmacology trials that NPL insulin has an action profile comparable to NPH insulin in subjects with type 1 diabetes. , However, a direct comparison of pharmacodynamic properties of insulin detemir and NPL insulin has not been performed to date.

To get further insight into the pharmacodynamic properties of insulin detemir compared with NPL insulin, this trial has been designed to compare pharmacodynamics in general and duration of action in particular between insulin detemir and NPL insulin in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
Primary objective:

The primary objective is to compare the pharmacodynamic response of insulin detemir and NPL insulin with respect to duration of action in a 32-hour euglycaemic glucose clamp experiment following single dose administration in subjects with type 1 diabetes.

Secondary objectives:

The secondary objectives are:

* to additionally characterise the pharmacodynamic profiles of insulin detemir and NPL insulin in a 32-hour euglycaemic glucose clamp experiment following single dose administration in subjects with type 1 diabetes.
* to characterise the pharmacokinetic profiles of insulin detemir and NPL insulin following single dose administration in subjects with type 1 diabetes.
* to assess the safety and tolerability of insulin detemir and NPL insulin following single dose administration in subjects with type 1 diabetes.

Trial design:

This is a randomised, single centre, double-blind, two-period crossover trial. Each subject will be randomly allocated to two single dose administrations on two separate dosing visits.

Trial population:

Thirty (30) male and female subjects with type 1 diabetes [age 18-65 years (incl.) and body mass index between 18.0 and 32.0 kg/m2 (incl.)] will be randomised into the trial.

Assessments:

Pharmacodynamics: The glucose infusion rate and plasma glucose concentration will be measured during a euglycaemic glucose clamp running for 32 hours after dosing.

Pharmacokinetics: Serum concentrations of insulin detemir and insulin lispro will be measured frequently during the first 32 hours after dosing.

Safety: Adverse events, laboratory safety variables (haematology, biochemistry, urinalysis), physical examination, vital signs and hypoglycaemic episodes.

Trial products:

* Insulin detemir (Levemir® Novo Nordisk), 100 U/mL in 3 mL Penfill® cartridges
* Insulin lispro protamine suspension (Humalog® NPL, Eli Lilly), 100 U/mL in 3 mL cartridges

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities.
2. Diagnosed with type 1 diabetes and treated with insulin
3. Male or female subject between 18 and 65 years of age
4. Body mass index between 18.0 and 32.0 kg/m2
5. HbA1c (glycosylated haemoglobin A1c) ≤ 11%
6. Fasting C-peptide ≤ 0.05 nmol/L
7. Treatment with intensified insulin therapy or continuous subcutaneous human insulin or insulin analogue infusion (CSII)] for at least 3 months.

Exclusion criteria

1. Known or suspected allergy to the trial products or related products,
2. Previous participation (randomised) in this trial.
3. The receipt of any investigational product within 3 months prior
4. Clinically significant abnormal haematology or biochemistry screening tests
5. Subject who is known to have hepatitis or who is a carrier of the Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies, or has a positive result to the test for HIV antibodies.
6. Supine blood pressure at screening (after 5 min in the supine position) ≥ 180 mmHg for systolic and/or ≥ 100 mmHg for diastolic. This exclusion criterion also pertains to subjects being on antihypertensives.
7. Clinically significant abnormal ECG at screening
8. Subject who has donated blood in excess of 500 mL within the 9 weeks preceding screening.
9. Significant history of alcoholism or drug/chemical abuse
10. Smoker
11. Subject with mental incapacity or language barriers
12. Surgery or trauma with significant blood loss within the 9 weeks preceding screening.
13. Subject with a history of or presence of cancer
14. History of any illness or disease that, in the opinion of the Investigator might confound the results of the trial or pose additional risk in administering the trial product to the subject.
15. Current systemic treatment with drugs that could interfere with glucose metabolism [such as systemic corticoids and monoamine oxidase (MAO) inhibitors] and/or pharmacokinetics.
16. Subject who has proliferative retinopathy or maculopathy and/or severe neuropathy (in particular autonomic neuropathy)
17. Any condition that would interfere with trial participation or evaluation of results, as judged by the Investigator and/or the sponsor.
18. Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Duration of action, time from onset of action until end of action | 32 h

SECONDARY OUTCOMES:
GIRmax, maximum glucose infusion AUCGIR,0-32h, AUCGIR,0-12h, AUCGIR,12-32h, tinf=0, Cmax,ins, tmax,ins, AUCins,0-24h AUCins,0-∞ AUCins,0-12h AUCins,12-24h | 0-32 h, 0-12 h, 0-24 h

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Study Director — Medical University Graz, Internal Medicine, Endocrinology and Nuclear Medicine
Locations (1):
- Medical University Graz, Graz, Graz, Austria